CLINICAL TRIAL: NCT06379373
Title: Peripheral Mechanisms of Humoral Immune Effector-mediated Tourette's Syndrome and the Role of Tuina Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-KLS-190-02
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Tourette Syndrome in Children; Food Intolerance; Inflammatory Response
Keywords: Tuina; Tourette Syndrome; Immune effectors; Mechanism
MeSH Terms: conditions — Food Intolerance; Tourette Syndrome | interventions — Manipulation, Spinal

STUDY DESIGN:
Intervention Model Description: According to the order of enrollment, the random number table method was used to divide the massage spinal manipulation+ placebo group (oral placebo, each dose: 50mg/time for 4-7 years old, 75mg/time for 7-12 years old, 100mg/time for 10-18 years old, 2 times/d), relaxation manipulation+ western medicine group (oral Typride tablets, each dose: 50mg/time for 4-7 years old, 75mg/time for 7-12 years old, 100mg/time for 10-18 years old, 2 times/d) for 2 consecutive weeks. Both groups were intervened for 2 courses. The observation time points were 2 weeks, 4 weeks, and 3 months before treatment and after treatment.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spinal manipulation (Experimental): Tuina method：(1) Cervical traction treatment (2) Relaxation techniques: Massage the neck for about 10 minutes with methods such as kneading, etc.
  (3) Orthopedic manipulation; (4) Cervicothoracic dorsal extension and wrenching method; (5) Lumbar spine oblique wrenching method;
  Interventions: Other: Spine manipulation; westren medicine
- Relaxation manipulation and medicine (Active Comparator): Take Typride tablets (Jiangsu Enhua Pharmaceutical Co., Ltd., Guoyao Zhunzi H32025477). Methods: Oral administration half an hour after meals. Dosage: 50mg/time for 4-7 years old, 75mg/time for 7-12 years old, 100mg/time for 10-18 years old, 2 times/d) for 23 cases each, 2 consecutive weeks for 1 course of treatment.
  Interventions: Other: Spine manipulation; westren medicine
- Healthy controls (No Intervention): healthy people

INTERVENTIONS:
Other: Spine manipulation; westren medicine — First Cervical traction,than spine release method,Massage the neck for about 10 minutes to realease muscles.Doctor use his two hands work together to pull the neck forward and upward,meanwhile, the patient's head is passively rotated to the right to the maximum, being rotated slightly with appropriate force, Doctor's left thumb pushes the crooked spinous process to the right, and the reduction sound can be heard at this time.
  If patient has upper thoracic spine misalignment, the dislocated segment needs to be adjusted.
  If patient has scoliosis, the affected spine segment should also be adjusted. If patient's lumbar facet joints are misaligned, or one of the lumbar muscles is spasmal, also the disorder joints need to be adjusted.
  Arms: Relaxation manipulation and medicine; Spinal manipulation

SUMMARY:
Tourette syndrome is a refractory type of tic disorder. Previous clinical studies have confirmed that Tuina has a good effect on TS, but the mechanism of action is still uncertain. Studies have found that the pathogenesis of TS may be related to immune factors, and patients will accompanied by the overflow of inflammatory factors such as interleukin-1β (IL-1β), interleukin-6 (IL-6), and tumor necrosis factor-α (TNF-α) during the onset of the disease. Other studies have found that the serum levels of IgG1, IgG2, IgG3, IgG4, IgGM, IgGA, IgGE, complement C3 and complement C4 are closely related to the pathogenesis of TS, and the abnormal humoral immune response mediated by food intolerance has an important impact on the pathogenesis of mental illness in children. The immune system plays a very complex role in TS. Based on this, we hypothesized that there may be differences in serum humoral immune effector levels between children with TS and healthy children, whether these differences are related to the consumption of certain allergenic foods or not, and so does Tuina spinal balancing can improve the clinical symptoms of children with TS by changing the levels of inflammatory and immune factors in peripheral serum. This study studied the peripheral mechanism of humoral immune effector mediated by Tourette syndrome and the intervention effect of Tuina through comprehensive scale analysis and advanced laboratory technology, which will provide a scientific theoretical basis and a safe and effective method for the treatment of multiple tics, and will have broad application prospects.

DETAILED DESCRIPTION:
1. Evaluation of TS clinical efficacy According to the Yale Tourette's Syndrome Global Severity Scale (YGTSS), the change in clinical control and the improvement rate of YGTSS score and TCM pattern score were evaluated. To investigate the changes in the clinical symptoms of children with TS before and after the intervention of Tuina Spinal Balance Method, and to confirm the effectiveness of this technique.
2. Serum interleukin-1β (IL-1β), interleukin-6 (IL-6), tumor necrosis factor-α (TNF-α) detection The levels of cytokines IL-1β, IL-6 and TNF-α in serum were detected by double-antibody sandwich enzyme-linked immunosorbent immunosorbent assay (ABS-ELSIA). To analyze the effect of Tuina spinal balancing method on inflammatory response in children with TS.
3. Quantitative immunoglobulin assays (1) Serum immunoglobulin IgG, IgM, IgA, IgE and IgG subclasses (IgG-1, IgG-2, IgG-3 and IgG-4) and complement C3 and complement C4 were detected by scattering turbidimetry. To analyze the response of Tuina spinal balancing method to humoral immunity in children with TS.

(2) The food-specific IgG4 and IgE detection kit provided by Beijing Deshankang Technology Co., Ltd. was used to test the serum IgG4 and IgE concentrations of the children by enzyme-linked immunoassay. After food-specific IgG4 and IgE analysis, the distribution of the positive rate of common food intolerance in children with TS was statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who meet the diagnostic criteria for TS；
* Haven't taken any drugs that affect the efficacy evaluation, such as antipsychotic drugs or traditional Chinese medicines with similar effects, or have received treatment but have passed the drug washout period for more than 1 month before enrollment；
* The legal guardian and the subject themselves have been informed consent, and have signed the informed consent form, agreeing to participate in this trial, and have been reviewed and approved by the Ethics Committee of Zhejiang Provincial Hospital of Traditional Chinese Medicine.

Exclusion Criteria:

* Any chorenia, Wilson's disease, epileptic myoclonus, drug-induced extrapyramidal symptoms and other extrapyramidal diseases;
* A history of severe tics;
* Any primary diseases such as cardiovascular, hepatic, renal and hematopoietic systems;
* Allergic or allergic to the drug in this test;
* Current taking other drugs or accept other treatments at the same time affect the evaluation of efficacy

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in scores on Yale global Tic severity scale(YGTSS) at Week4 and Week8 | Baseline and Week4 and Week8
  These include motor tics, vocal tics, and social impairment scores. Among them, motor and vocal tics were divided into five items: type of tic, frequency, intensity, complexity and interference, each item was recorded as 0, 1, 2, 3, 4 and 5 points. According to the severity, the higher score is , the more severe the severity represent. In order of severity, they are scored as 0 (no effect), 10 (little difficulty), 20 (minor difficulty), 30 (significant difficulty), 40 (fairly difficult) and 50 (very difficult).The sum of motor tics score + vocal tic score + social impairment score is recorded as the total Yale score.
Change from Baseline in scores on TCM Syndrome Points at Week4 and Week8 | Baseline and Week4 and Week8
  The scale includes 5 main symptoms, including frowning or blinking, opening or grinning, shaking or shrugging shoulders, shaking hands or kicking, speaking in different or obscene words, muscle twitches, yellow face or emaciation or obesity, mental fatigue or loss of appetite, difficulty concentrating or forgetfulness and insomnia, irritable temperament or temper or difficulty sitting still or restlessness at night, irregular bowel movements, tongue and pulse.
  The main symptoms are scored 0, 1, 2, 3 and 4 points according to the symptoms from mild to moderate, and the secondary symptoms are scored 0, 1 and 2 points respectively according to the symptoms from mild to severe. Tongue quality (pale red 0 points, red 1 point, red 2 points). Tongue coating (0 points for moss peeling, 1 point for moss thin white, 2 points for moss white and greasy), pulse (0 points for peace, 2 points for fine/fine strings).

SECONDARY OUTCOMES:
Change from Baseline in difference in the spacing of the lantoine side | Baseline and Week4 and Week8
  According to X-ray mouth opening images of the child before and after treatment between two groups

CONTACTS AND LOCATIONS:
Overall Officials: xiaojuan Li, Principal Investigator — The First Affiliated Hospital of Zhejiang Chinese Medical University
Locations (1):
- First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No